CLINICAL TRIAL: NCT03197610
Title: The Effect of Enamel Matrix Derivatives on Root Coverage Esthetic Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hacer Sahin Aydinyurt, Assistant professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.YYU.0.01.00.0
Record Dates: First submitted 2017-06-15; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Gingival Recession; Periodontal Diseases
Keywords: gingival recession; sub epithelial connective tissue graft; enamel matrix derivatives; root coverage aesthetic score
MeSH Terms: conditions — Gingival Recession; Periodontal Diseases | interventions — enamel matrix proteins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCTG+EMD (Experimental): TEST GROUP: Langer and Langer technique was used to prepare the recipient side. The vestibule surfaces of adjacent interdental papillae were de-epithelialized. The dimensions of the recipient area were measured by periodontal probes and four bleeding centers were created in the palatinal region. The graft was placed on the recipient site and fixed with 4.0 silk sutures. Pressure was applied to the operation area for 5 minutes with saline impregnated sponges. EMD (Emdogain®, Straumann, Basel, Switzerland) was used in the test group in addition to SCTG. Prior to EMD application, the root surface was applied with 24% EDTA (PrefGel, Straumann, Basel, Switzerland) for 2 minutes. The area was washed with saline and then EMD was applied.
  Interventions: Procedure: enamel matrix derivatives
- ONLY SCTG (Experimental): CONTROL GROUP: Langer and Langer technique was used to prepare the recipient side. The anesthetic solution was applied to the donor site in the palatinal region on the same side as the operation site. The dimensions of the recipient area were measured by periodontal probes and four bleeding centers were created in the palatinal region. The graft was placed on the recipient site and fixed with 4.0 silk sutures. Pressure was applied to the operation area for 5 minutes with saline impregnated sponges.
  Interventions: Procedure: enamel matrix derivatives

INTERVENTIONS:
Procedure: enamel matrix derivatives — enamel matrix derivatives and subepithelial connective tissue grafts

SUMMARY:
Subepithelial connective tissue grafts (SCTG) are accepted as the gold standard in covering denuded root surfaces. Combining enamel matrix derivatives (EMD) with periodontoplasic surgical operations is another method in covering denuded root surface. The aim of this study is to compare a SCTG operation group and EMD applied group in addition to SCTG using complete root coverage rate and a newer method root coverage esthetic scoring system (RES).

DETAILED DESCRIPTION:
Background: Subepithelial connective tissue grafts (SCTG) are accepted as the gold standard in covering denuded root surfaces. Combining enamel matrix derivatives (EMD) with periodontoplasic surgical operations is another method in covering denuded root surface. The aim of this study is to compare a SCTG operation group and EMD applied group in addition to SCTG using complete root coverage rate and a newer method root coverage esthetic scoring system (RES).

Methods: This is a split-mouth and controlled study. Thirthy-eight Class I or II gingival recession defects at canine teeth were treated in the control (SCTG) (n=19) and test groups (n=19) (SCTG+EMD). The root coverage esthetic score were evaluated by 2 blind periodontists 1 year after the treatment using RES. The agreement between the two periodontists was assessed by kappa analysis. Complete root coverage rate was evaluated for both groups. Two groups were compared with statistically methods in terms of RES parameters and gingival recession height /width.

ELIGIBILITY:
Inclusion Criteria:

* The patient had no systemic disease, did not smoke cigarette and tobacco products, did not have a pregnancy and breastfeeding period, had class I and class II gingival recession according to the Miller gingival classification, had a recession depth of ≥2 mm, have not had a restoration and have had an operation in the relevant dental region that had no previous gingival surgical procedure were included in this study.

Exclusion Criteria:

* systemic disease
* multiple gingival recession
* miller class III and IV recessions were excluded

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
root coverage percentage | 1 year
  root coverage percentage of denuded root surface
root coverage aesthetic score | 1 year
  root coverage aesthetic score of treatment modalities

IPD SHARING:
Plan to Share IPD: Yes